CLINICAL TRIAL: NCT01802528
Title: Clinical Effectiveness of Obturator Externus Muscle Injection in Chronic Pelvic Pain Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0924
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Pelvic Pain
Keywords: obturator externus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obturator externus muscle injection: patients were treated with obturator externus injection

SUMMARY:
Obturator externus (OE) muscle has the possibility as a pain generator, considering its anatomical and functional aspects, but this muscle as a possible target for therapeutic intervention is currently understudied in pain practice.

ELIGIBILITY:
Inclusion Criteria:

* 1. 20-75 adults/ 2. Chronic pelvic pain patients who required the interventional procedures/ 3. patients with a localized tenderness on inferolateral side of the pubic tubercle

Exclusion Criteria:

* 1. Severe cardiovascular disease /2. Coagulation abnormality /3. Patient denial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was defined as chronic pelvic pain patients with a localized tenderness on inferolateral side of the pubic tubercle corresponding to obturator foramen who received OE muscle injection with local anesthetic for their pain treatment.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Post-injection pain score | at 2 weeks after injection
  Before and after the OE muscle injection, patients were asked to rate their pain score using a 10-point numeric rating scale (NRS; 0=no pain, 10=worst possible pain). We also assessed the degree of patient satisfaction as excellent, good, fair, and bad during 2 weeks after injection. In this period, any analgesic medications did not change in all patients. Complications associated with OE muscle injection were investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute,, Seoul, Seoul, South Korea